CLINICAL TRIAL: NCT02853552
Title: Use of Misoprostol by Families and Women as a First Aid Measure to Address Excessive Postpartum Bleeding in Home Deliveries
Brief Title: Misoprostol as First Aid Measure to Address Excessive Postpartum Bleeding
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Gynuity Health Projects (Other)
Collaborators: National Committee for Maternal & Neonatal Health (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 3007
Record Dates: First submitted 2016-07-29; First posted 2016-08-03 (Estimated); Last update posted 2016-08-03 (Estimated); Status verified 2016-07

CONDITIONS: Postpartum Hemorrhage
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — Misoprostol

INTERVENTIONS:
Drug: Misoprostol — 800mcg misoprostol taken sublingually

SUMMARY:
The overall study purpose is to evaluate the safety, feasibility and acceptability of advance distribution of misoprostol to be used as 'first aid treatment' administered by the woman herself or her family to help treat excessive bleeding in home births.

DETAILED DESCRIPTION:
This is a quasi-experimental, pre-post intervention study that will be conducted over a period of 12 months and will span two phases:

Phase 1 (baseline) (6 months): Data on deliveries will be collected for pregnant women who deliver during this phase. Data will also be collected on the treatment administered in any PPH cases. Women will be counseled on and also receive educational materials on how to identify excessive bleeding and the importance of seeking care at a facility if excessive bleeding occurs.

Phase 2 (misoprostol) (6 months): During this phase, the study will pilot the first aid concept. Women will be provided with a single dose of 800 mcg sublingual misoprostol (200 mcg x 4 tablets) during their third trimester to use in the event of excessive postpartum bleeding, as well as the educational materials and counseling provided during the Phase 1. The misoprostol is intended to serve as a first aid treatment measure and although seeking additional care is challenging in this setting, women and families will be advised to have a plan ready to seek immediate care at a health facility as soon as they take the misoprostol.

During both study phases, data will be collected on maternal, clinical, and neonatal outcomes for all deliveries that occur in the study area. If women receive any care related to their delivery, data collectors will document this information.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women living in sample districts

Exclusion Criteria:

* Unable to provide informed consent

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 4330 (Estimated)
Dates: Start 2016-10; Primary Completion 2017-10 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Number of cases identified as having excessive bleeding | Within 1 week after delivery
Proportion of women who administer misoprostol as first aid | Within 1 week after delivery
  Proportion of women who took misoprostol to treat excessive bleeding out of women who self-diagnosed excessive bleeding
Proportion of women who correctly administer misoprostol as first aid | Within 1 week after delivery
  Proportion of women who administer misoprostol by correct route and correct dose for treatment of excessive bleeding out of all women who administer misoprostol for treatment of excessive bleeding
Acceptability of side effects of misoprostol | Within 1 week after delivery
Number of women who are transferred for excessive bleeding | Within 1 week after delivery
  Women who are receive care for heavy bleeding by a skilled provider at home or at a health facility
Proportion of women who experience a serious adverse event due to excessive bleeding | Within 1 week after delivery
  Proportion of women who experience a SAE (defined as laparotomy, surgery, hysterectomy, blood transfusion or death) out of all women who experience excessive bleeding
Proportion of women who receive an additional intervention (e.g. use of additional uterotonic or suturing) for excessive bleeding | Within 1 week after delivery
Level of acceptability and satisfaction with using misoprostol as first-aid option to treat excessive bleeding | Within 1 week after delivery
Correct comprehension of information related to misoprostol and its use for first aid | Within 1 week after delivery
  Proportion of women who correctly answer questions related to use and administration of misoprostol for first aid to treat excessive bleeding

IPD SHARING:
Plan to Share IPD: No